CLINICAL TRIAL: NCT03575598
Title: Sitravatinib (MGCD516) and Nivolumab in Oral Cavity Cancer Window Opportunity Study (SNOW)
Brief Title: Sitravatinib (MGCD516) and Nivolumab in Oral Cavity Cancer Window Opportunity Study
Acronym: SNOW
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNOW-001
Record Dates: First submitted 2018-06-11; First posted 2018-07-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Squamous Cell Carcinoma, Head And Neck; Squamous Cell Carcinoma Mouth; Squamous Cell Carcinoma of the Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — sitravatinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sitravatinib and Nivolumab (Experimental): Patients will start therapy with sitravatinib within 10 days of study enrollment. Sitravatinib will be given at 120mg once daily on a continuous basis until 48 hours before planned surgery, or for a maximum period of 28 days.
  Nivolumab will be given as a single infusion at a dose of 240mg, over a period of 30 minutes on Day 15 of the study.
  Interventions: Drug: Sitravatinib; Biological: Nivolumab

INTERVENTIONS:
Drug: Sitravatinib — Sitravatinib (MGCD516) is an orally-available, potent small molecule inhibitor of a closely related spectrum of tyrosine kinases, which has shown antitumor activity in a variety of in vitro and in vivo model systems.
  Other Names: MGCD516
Biological: Nivolumab — Nivolumab (OPDIVO®) is a human IgG4 kappa immunoglobulin that binds to the PD-1 receptor and blocks its interaction with PD-L1 and PD-L2, releasing PD-1 pathway-mediated inhibition of the immune response, including the anti-tumor immune response.
  Other Names: OPDIVO®

SUMMARY:
This is a window of opportunity study for patients with resectable squamous cell carcinoma of the oral cavity who are considered suitable for curative-intent surgical resection, with pre-operative drugs, Sitravatinib and Nivolumab.

DETAILED DESCRIPTION:
This is a single center, open-label, non-randomized, pre-operative window of opportunity study for patients with resectable squamous cell carcinoma of the oral cavity who are considered suitable for curative-intent surgical resection, with pre-operative Sitravatinib and Nivolumab. A total of 12 patients who are evaluable for correlative studies, are planned for enrollment.

This study will involve treatment with Sitravatinib and Nivolumab, tests and procedures done for safety and the collection of blood samples for biomarker research. Tissue samples (fresh biopsy or archival tissue) will also be collected for biomarker research and evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written and voluntary informed consent.
2. Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
3. Age > 18 years, male or female.
4. Patient must be diagnosed with histologically confirmed squamous cell carcinoma of the oral cavity (SCCOC) (floor of mouth, anterior 2/3 tongue, buccal mucosa, upper and lower gingiva, retromolar trigone and hard palate) previously untreated, considered resectable by the head and neck treating surgeon (T2-4a, N0-2, or T1 - greater than 1 cm - N2, M0; without evidence of distant metastasis).
5. Patient must be willing and able to provide 2 fresh tumor biopsies for histopathological and biomarker evaluation: one at baseline and one after treatment with Sitravatinib but prior to treatment with Nivolumab. Archival tissue sample will be requested if available.
6. No anti-neoplastic treatment is allowed between the time from obtaining baseline tumor specimen and enrollment.
7. ECOG performance status 0-1.
8. Patient must have adequate organ function as determined by the following:

   • Renal function: i. Serum creatinine < 1.5 ULN (upper limit of normal range) or a calculated creatinine clearance of > 50mL/min using the following formula:

   Creatinine clearance = [(140-age) x wt (kg) x Constant*] / creatinine (umol/L)

   *Constant = 1.23 for men, and 1.04 for women

   • Bone marrow function (without hematopoietic growth factors or transfusion): i. Absolute neutrophil count (ANC) > 1.0 x 109/L ii. Leukocytes > 2.0 x 109/L iii. Hemoglobin > 90 g/L or > 9g/dL iv. Platelets > 100 x 109/L

   • Liver function: i. Total bilirubin ≤ 1.5 x ULN or ≤ 3 x ULN for patients with Gilbert Syndrome. ii. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) < 2.5 x ULN

   • Cardiac function: i. A normal left ventricular ejection fraction (LVEF) of ≥50% by a MUGA scan performed within 4 weeks of the study commencement.
9. Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy). Women of child-bearing potential (WOCBP) or men whose partner is a WOCBP agrees to use contraception while participating in this study, and for a period of 6 months following termination of study treatment.
10. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Primary site of head and neck carcinoma unknown, lip, skin, or outside the oral cavity.

   • Patients with tumors that invade major vessels or are within ≤ 3 mm of the carotid artery as shown unequivocally by imaging studies.
2. Patients with any prior history of clinically significant bleeding related to the current head and neck cancer.
3. Patients with a history of gross hemoptysis (bright red blood of ½ teaspoon or more per episode of coughing) < 3 months prior to enrollment.
4. Prior or concurrent radiation therapy to tumor at site of planned resection.
5. Any concurrent chemotherapy, biologic, immunologic or hormonal therapy for cancer treatment.

   • Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
6. Current or prior use of immunosuppressive medication within 14 days prior to starting dosing. The following are exceptions to this criteria:

   * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection).
   * Adrenal replacement steroid > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
   * Steroids as premedication for hypersensitivity reactions (eg, computed tomography scan premedication).
7. Active or documented history of autoimmune disease within 2 years before screening, including:

   * Active or prior documented inflammatory bowel disease (eg. Crohn's disease, ulcerative colitis).
   * Patients with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, Grave's disease, Hashimoto's disease, or psoriasis not requiring systemic steroids and/or immunosuppressive agents within the past 2 years, are not excluded.
8. History of primary immune deficiency.
9. History of stroke or transient ischemic attack within the previous 6 months.
10. History of uncontrolled hypertension (> 150 mm Hg systolic or > 100 mm Hg diastolic) on multiple observations despite standard of care treatment.
11. Any of the following cardiac abnormalities:

    * Unstable angina pectoris,
    * Congestive heart failure ≥ NYHA Class 3,
    * QTc >480 milliseconds,
    * Left ventricular ejection fraction (LVEF) < 50.
12. Concomitant medication known to cause prolonged QT that cannot be discontinued or changed to a different medication prior to enrollment.
13. History of organ transplant that requires use of immunosuppressive medications.
14. Known allergy or reaction to any components of Sitravatinib and/or Nivolumab formulation.
15. Subjects who are known to be human immunodeficiency (HIV) positive.
16. Has a known history of or is positive for active hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (defined as HCV RNA [qualitative] is detected).

    * HBV DNA must be undetectable and HBsAg negative at Screening Visit.
    * Participants who have had definitive treatment for HCV are permitted if HCV RNA is undetectable at Screening Visit.
17. Female patients who are pregnant or breast-feeding.
18. Uncontrolled intercurrent illness including, but not limited to, ongoing or active clinically significant infection requiring parenteral antibiotics, unstable cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events from Sitravatinib or Nivolumab, or compromise the ability of the subject to give written informed consent.
19. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study regimen or interpretation of patient safety or study results.
20. Any previous treatment with a PD1 or PD-L1 inhibitor, including Nivolumab.
21. History of another primary malignancy, except for:

    * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence,
    * Adequately treated non-melanoma skin cancer without evidence of disease,
    * Adequately treated carcinoma in situ without evidence of disease.
22. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study medications.
23. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic and immune effects of pre-operative therapy with Sitravatinib and Nivolumab in patients with SCCOC | 2 years
  Tumor PD-L1 expression by IHC
Pharmacodynamic and immune effects of pre-operative therapy with Sitravatinib and Nivolumab in patients with SCCOC | 2 years
  Density of immune cell population in the tumor and/or peripheral blood, including circulating tumor DNA (ctDNA), T-cell subsets, NK cells and myeloid-derived cell subsets
Pharmacodynamic and immune effects of pre-operative therapy with Sitravatinib and Nivolumab in patients with SCCOC | 2 years
  Serum pro-inflammatory cytokines and chemokines

SECONDARY OUTCOMES:
Safety and tolerability of pre-operative therapy with Sitravatinib and Nivolumab on patients with SCCOC | 2 years
  Toxicities as per NCI CTCAE v5.0
Safety and tolerability of pre-operative therapy with Sitravatinib and Nivolumab on patients with SCCOC | 2 years
  Rate of completion of surgery within the initially planned window
Safety and tolerability of pre-operative therapy with Sitravatinib and Nivolumab on patients with SCCOC | 2 years
  Rate of post-operative complications
Pre-operative clinical activity of the combination of Sitravatinib and Nivolumab in patients with SCCOC | 2 years
  Rate of disease progression as per RECIST v1.1 during the pre-operative treatment period
Pre-operative clinical activity of the combination of Sitravatinib and Nivolumab in patients with SCCOC | 2 years
  Pathologic treatment effect in tumor and/ or lymph nodes
Pre-operative clinical activity of the combination of Sitravatinib and Nivolumab in patients with SCCOC | 2 years
  Rate of nodal extracapsular extension and positive margins
Sitravatinib plasma levels alone and in combination with Nivolumab. | 2 years
  Analysis of plasma Sitravatinib concentration before and after Nivolumab therapy

OTHER OUTCOMES:
Dynamic changes in immune cell activation and/or suppression using flow cytometry, DNA/RNA sequencing, and FACS sorting | 2 years
  Additional tumor cell surface marker expression
Dynamic changes in immune cell activation and/or suppression using flow cytometry, DNA/RNA sequencing, and FACS sorting | 2 years
  Flow cytometry analysis of activation markers on circulating immune cells
Dynamic changes in immune cell activation and/or suppression using flow cytometry, DNA/RNA sequencing, and FACS sorting | 2 years
  Tumor and immune cell genome and transcriptome analysis
Dynamic changes in intratumoral hypoxia with pre-operative Sitravatinib and Nivolumab therapy | 2 years
  Analysis of tumor 18FAZA-PET uptake patterns

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliva M, Chepeha D, Araujo DV, Diaz-Mejia JJ, Olson P, Prawira A, Spreafico A, Bratman SV, Shek T, de Almeida J, R Hansen A, Hope A, Goldstein D, Weinreb I, Smith S, Perez-Ordonez B, Irish J, Torti D, Bruce JP, Wang BX, Fortuna A, Pugh TJ, Der-Torossian H, Shazer R, Attanasio N, Au Q, Tin A, Feeney J, Sethi H, Aleshin A, Chen I, Siu L. Antitumor immune effects of preoperative sitravatinib and nivolumab in oral cavity cancer: SNOW window-of-opportunity study. J Immunother Cancer. 2021 Oct;9(10):e003476. doi: 10.1136/jitc-2021-003476. PMID 34599023